CLINICAL TRIAL: NCT01028430
Title: B Cell Repertoires in Chronic Lymphocytic Leukemia and Aging
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 04-046
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Blood cells, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia: Chronic Lymphocytic Leukemia

SUMMARY:
B-CLL is the most prevalent leukemia in the Western hemisphere, accounting for ~25% of all leukemia's (1). This disease occurs virtually exclusively in the aging population, with the median age of diagnosis ranging between the mid 60s and the early 70s. Indeed, its occurrence before the age of 50 is quite unusual. This increase in occurrence with age is not unique to B-CLL; rather, it is characteristic several B cell lymphoproliferative disorders (e.g., non-Hodgkin's lymphoma, multiple myeloma). Gender and race also influence the development of B-CLL. Thus, the ratio of men: women is ~2:1 and the prevalence is increased in Caucasians. The rate of occurrence of B-CLL among Asians is significantly lower than for Caucasians and this does not increase with immigration to the West. DNA sequence analyses performed in our laboratory and in those of others indicate that B-CLL cells from unrelated patients share Ig V gene characteristics. These include the use of selected genes, the association of these genes with certain D and JH gene segments that code for unique CDR3 motifs, and the occasional occurrence of highly similar VHDJH + VLJL pairs. In ~50% cases, these rearranged genes are mutated, whereas in the others mutations are infrequent; this difference is related to the VH gene family used by the B-CLL cell.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age Patients must be willing to be contacted in the future

Exclusion Criteria:

* Patients who are known to be anemic, with a hemoglobin <8 PAtients who are known to be infected with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Lymphocytic Leukemia Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 1998-07; Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
expression of cell surface antigens HLA-DR and CD38+ markers in B-CLL cells compared to normal B-lymphocytes | samples will be taken at the beginning, week 2, 4,6,8,12,and 24 (for blood), and bone marrow samples at weeks 2 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Chiorazzi, MD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States